CLINICAL TRIAL: NCT05487794
Title: Effect of Dose Fractionation of Testosterone Cypionate on Hematocrit in Transgender Men with Erythrocytosis Secondary to Testosterone Use.
Brief Title: Effect of Dose Fractionation of Testosterone Cypionate on Transgender Men with Erythrocytosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, SERGIO HENRIQUE PIRES OKANO, Principal investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DGO-777
Record Dates: First submitted 2022-07-26; First posted 2022-08-04 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Testosterone; Transsexualism; Hematologic Diseases
MeSH Terms: conditions — Transsexualism; Hematologic Diseases | interventions — testosterone 17 beta-cypionate

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (T100) (Experimental)
  Interventions: Drug: Testosterone Cypionate 100 MG/ML
- Group 1 (T0) (No Intervention)

INTERVENTIONS:
Drug: Testosterone Cypionate 100 MG/ML — Testosterone is also responsible for increasing hematocrit by stimulating erythropoiesis (Velho et al., 2017). In cisgender men, who are hypogonadal and do not adequately produce testosterone, treatment with the use of testosterone is associated with stimulation of erythropoiesis, which can potentially increase blood viscosity, resulting in secondary erythrocytosis (Hajjar et al., 1997).
  Arms: Group 1 (T100)

SUMMARY:
A transgender man is someone with a male identity who were born with a vulva and vagina. The acquisition of masculine characters can come from surgery or from the use of testosterone. Despite the benefit of using this hormone in relation to hair development, muscle mass gain and changes in voice timbre, its use can cause an increase in the hematocrit (Ht) level. When erythrocytosis occurs (Ht ≥ 50%), the currently proposed conduct is the suspension of cross-hormonization for 3 months, which has negative effects on the affirmation process. This project aims to assess whether reducing the dose of testosterone cypionate by half (100mg/15d) can mitigate the negative outcomes caused by the suspension with the benefit of reducing the hematocrit level in trans patients who developed erythrocytosis using testosterone. This is a pilot study that will compare the intervention (testosterone cypionate 100 mg, fortnightly) to the suspension of the drug, both for 3 months, with the main outcome being the hematocrit level. Hormonal and biochemical levels and the Hospital Anxiety and Depression scale (HAD) will also be evaluated in patients treated at the Gender Incongruence Outpatient Clinic of the Hospital das Clínicas of the Faculty of Medicine of Ribeirão Preto.

ELIGIBILITY:
Inclusion Criteria:

* TM aged between 18 and 40 years in threatmeant with Testosterone Cypionate 200mg/2mL with a diagnosis of erythrocytosis (Ht⩾50%).

Exclusion Criteria:

* TM with polycythemia vera or secondary to other pathologies (chronic kidney disease, severe lung disease, chronic myeloid leukemia, lymphoma, liver diseases and Cushing's syndrome);
* TM in use of hormonal contraceptives or copper IUDs;
* TM with psychiatric conditions such as severe psychotic disorders, severe personality disorders
* Patients with Ht > 54.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male transgender
Enrollment: 46 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Rate of Erythrocytosis | 3 months
  To evaluate if the reduction of the dose of Testosterone Cypionate 200 mg to 100 mgm, biweekly, is effective to normalize the hematocrit in TM with erythrocytosis. Hemoglobin and hematocrit: will be measured by automated counting in the Biochemistry laboratory of the HCRP, using the Siemens Advia 2120i device (Siemens Healthcare GmbH®, Munich, Germany). Blood collection will be carried out in Recrututo and 3 months after intervention or control.

SECONDARY OUTCOMES:
Efects on lipids and glucose levels | 3 monsths. Blood collection will be carried out in recruitment and 3 months after intervention or control.
  Blood samples will be collected between seven and eight in the morning, after a minimum of twelve hours fasting. In each evaluation, 20 mL of whole blood will be collected and stored in conical plastic tubes (BD-Becton Dickinson, Plymouth, United Kingdom) with a vacuum and a separating gel barrier. It will be measured: total cholesterol (TC), HDL-cholesterol and triglycerides (TG) by enzymatic method in the Biochemistry laboratory of HCRP. The device used will be the Siemens Atellica CH 930 (Siemens Healthcare GmbH®, Munich, Germany). LDL-cholesterol will be calculated from the Friedewald formula, if there is no dosage of TG greater than 400mg/dL (Friedewald et al., 1972). Fasting blood glucose will be determined by the enzymatic method in the Biochemistry laboratory of the HCRP and the device used will be the Siemens Atellica CH 930 (Siemens Healthcare GmbH®, Munich, Germany)
Anxiety and Depression Hospital Scale (HAD) | The scale will be applied in recruitment and 3 months after intervention or control.
  To evaluate the emotional state regarding the presence of anxiety and depression, the Brazilian version of the Hospital Anxiety and Depression Scale (HAD) will be used, which consists of 14 questions that assess some aspects of mood and behavior (Appendix 4). Scores ≥ 9 in the questions corresponding to anxiety or depression characterizes the psychic state of the woman.Zigmond & Snaith, 1983).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculdade de Medicina de Ribeirão Preto - FMRP-USP, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided